CLINICAL TRIAL: NCT04856345
Title: The Effect of a 4 Week Auditory-motor Coupling Intervention on Walking, Information Processing Speed and Fatigue in Persons With Multiple Sclerosis: Three Armed Pilot Intervention
Brief Title: Running Title: Walking to Music and in Silence on a Treadmill
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasselt University (Other)
Collaborators: Revalidatie & MS Centrum Overpelt (Other)
Responsible Party: Principal Investigator, Peter Feys, Principal Investigator, Hasselt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B1152020000021
Record Dates: First submitted 2021-02-02; First posted 2021-04-23 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Walking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Music with synchronising (Experimental): walking to music that one can synchronise to
  Interventions: Other: Walking with music with synchronisation
- Music without synchronising (Active Comparator): walking to music that one cannot synchronise to
  Interventions: Other: Walking with music without synchronisation
- No music (Sham Comparator): walking without music.
  Interventions: Other: walking without music

INTERVENTIONS:
Other: Walking with music with synchronisation — Walking with music than one can synch to
  Arms: Music with synchronising
Other: Walking with music without synchronisation — Walking with music than one cannot synch to
  Arms: Music without synchronising
Other: walking without music — Walking without music
  Arms: No music

SUMMARY:
This work is embedded in the context of auditory-motor coupling, which entails the engagement of two systems; the interaction between the music (or repetitive auditory stimuli) and a walking individual (repetitive movements of footfall). In previous studies, the investigators have shown that synchronising steps to beats in music have shown to be feasible in persons with multiple sclerosis, showing increase of step frequency and reduced perceived fatigue[1, 2]. In this current work, The investigators expand previous findings with a pilot intervention study, to investigate if synchronisation is necessary to improve cognitive and motor functions.

The proposed experiment includes 30 participants, randomised to three arms of a pilot intervention (10 participants per arm). With the intention of a further case-study analysis, the inestigators request to include 4 additional participants (2 PwMS with cognitive impairment, and 2 persons with cerebellar lesion) to only follow the intervention arm 1.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of MS if >1,
* no relapses >1 month,
* ability to walk for 12minutes,
* ability to walk independently on a treadmill
* walking speed between 0.8-1.2m/s.

Exclusion Criteria:

* amusia,
* deafness,
* cognitive impairment hindering understanding of study instructions,
* pregnancy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-01-22 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
12- item multiple sclerosis walking scale | Baseline
  The Multiple Sclerosis Walking Scale is a self-assessment scale which measures the impact of MS on walking. It consists of 12 questions concerning the limitations to walking due to MS during the past 2 weeks. Each item can be answered with 5 options, with 1 meaning no limitation and 5 extreme limitation.
12- item multiple sclerosis walking scale | week 5
  The Multiple Sclerosis Walking Scale is a self-assessment scale which measures the impact of MS on walking. It consists of 12 questions concerning the limitations to walking due to MS during the past 2 weeks. Each item can be answered with 5 options, with 1 meaning no limitation and 5 extreme limitation.
6 minutes walking test to calculate the distance walking Index | Baseline
  impact of MS on walking
6 minutes walking test to calculate the distance walking Index | week 5
  impact of MS on walking
12 minute walking with sensors | Baseline
  gait dynamics and pattern - detrended fluctuation analysis and spatio-temporal parameters
12 minute walking with sensors | week 5
  gait dynamics and pattern - detrended fluctuation analysis and spatio-temporal parameters

SECONDARY OUTCOMES:
Paced auditory serial addition test and symbol digit modality test | Baseline
  to measure cognitive functioning and cognitive fatigability
Paced auditory serial addition test and symbol digit modality test | week 5
  to measure cognitive functioning and cognitive fatigability
Motricity Index of dorsi flexors, knee extensors and hip flexors | Baseline
  Muscle weakness
Motricity Index of dorsi flexors, knee extensors and hip flexors | week 5
  Muscle weakness
Modified Aschowrth scale Hamstrings, Tricepts Surae, Quadricepts | Baseline
  Spasticity
Modified Aschowrth scale Hamstrings, Tricepts Surae, Quadricepts | week 5
  Spasticity
Scale for the assessment and rating of ataxia | Baseline
  Ataxia
Scale for the assessment and rating of ataxia | week 5
  Ataxia
Dynamic gait index | Baseline
  Dynamic balance
Dynamic gait index | week 5
  Dynamic balance
Time up and Go test | Baseline
  balance
Time up and Go test | week 5
  balance
Modified fatigue impact scale | Baseline
  self-reported outcomes for fatigue
Modified fatigue impact scale | week 5
  self-reported outcomes for fatigue
Barcelona music reward questionnaire | Baseline
  experience of music reward
Barcelona music reward questionnaire | week 5
  experience of music reward
Hospital anxiety and depression questionnaire | Baseline
  anxiety and depression
Hospital anxiety and depression questionnaire | week 5
  anxiety and depression
Activities-specific balance confidence scale | Baseline
  self-reported outcome for activity and balance
Activities-specific balance confidence scale | week 5
  self-reported outcome for activity and balance
Stroke rehabilitation motivation scale | Baseline
  self-reported motivation questionnaire
Stroke rehabilitation motivation scale | week 5
  self-reported motivation questionnaire
the Brunnel Music Rating Inventory-2 | Baseline
  self-reported music rating inventory
the Brunnel Music Rating Inventory-2 | week 5
  self-reported music rating inventory
credibility and expectations questionnaire | week 5
  self-reporting of credibility of the intervention.
Pre and Post training sessions, 2x a week, 20 minutes for 4 weeks | up to week 4
  Before and after each training session
  * Perceived cognitive and physical fatigue rated on a visual analogue scale
  * Perceived motivation rated on a Likert scale

CONTACTS AND LOCATIONS:
Overall Officials: Peter Feyse, prof. dr., Principal Investigator — Hasselt University; Lousin Moumdjian, dr., Study Chair — Hasselt University
Locations (1):
- Noorderhart Revalidatie & MS centrum, Overpelt, Belgium